CLINICAL TRIAL: NCT00410800
Title: Insulin Secretory Defects in Pima Indians at High Risk for NIDDM
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999996032; OH96-DK-N032
Record Dates: First submitted 2006-12-12; First posted 2006-12-13 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-08-16

CONDITIONS: NIDDM
Keywords: Insulin Resistance; Body Composition; Kinetic Modeling
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

SUMMARY:
The Pima Indians have the highest reported prevalence of NIDDM of any population in the world. Within this population, it is possible to identify subgroups of individuals at a particularly high risk for NIDDM. This project examines whether defects in insulin secretion contribute to the higher risk of NIDDM in these subgroups and whether they progress over the course of the disease.

Healthy Pima men and women at high risk for NIDDM including individuals in the following 3 groups will be recruited: 1)persons whose mothers and/or father developed diabetes at an early age (< 35 y); 2) persons whose mothers were diabetic during pregnancy; and 3) persons whose birthweight was < 2500 g. These individuals, as well as subjects with none of the above risk factors and a group of non-Pima controls, will be admitted to the NIH Clinical Research Unit at Phoenix Indian Medical Center for the following series of studies. Body composition will be determined by DXA scanning and by measuring the amount os visceral abdominal fat using MRI. A 75-g oral glucose tolerance test and a 25-g intravenous glucose tolerance test will be performed. Insulin action will be measured with a hyperinsulinemic-euglycemic glucose clamp (insulin infusion: 40mU/m(2) min and insulin secretory responses to glucose will be measured during a 5-step hyperglycemic glucose clamp immediately thereafter. Pima subjects will be followed longitudinally after discharge from the unit and oral glucose tolerance tests will be performed every three months. Individuals who transition from normal to impaired glucose tolerance or impaired glucose tolerance to diabetic will be invited back to the Clinical Research Center for repeat testing.

By comparing insulin secretion-glucose dose-response curves, it may be possible to discern subtle defects in insulin secretion predisposing certain individuals to NIDDM. In addition, comparison of the responses in the offspring of diabetic pregnancies with those in the offspring of mothers who subsequently became diabetic may allow us to separate defects due to genetic causes from those due to the intrauterine environment. Finally, studying subjects as they progress from normal glucose tolerance to diabetes will test whether the defects in insulin secretion are progressive and contribute to the development of NIDDM.

DETAILED DESCRIPTION:
The Pima Indians have the highest reported prevalence of NIDDM of any population in the world. Within this population, it is possible to identify subgroups of individuals at a particularly high risk for NIDDM. This project examines whether defects in insulin secretion contribute to the higher risk of NIDDM in these subgroups and whether they progress over the course of the disease.

Healthy Pima men and women at high risk for NIDDM, including individuals in the following 4 groups, will be recruited: 1) persons whose mother and/or father developed diabetes at an early age (less than 35 y); 2) persons whose mothers were diabetic during pregnancy; 3) persons whose birth-weight was less than 2500 g; and 4) persons with enlarged abdominal fat cells (greater than 1.08 microgram lipid/cell). These individuals, as well as subjects with none of the above risk factors and a group of non-Pima controls, will be admitted to the NIH Clinical Research Unit at Phoenix Indian Medical Center for the following series of studies. Body composition will be determined by DXA scanning and by measuring the amount of fat in the abdomen and thigh using MRI. Fat cell size will be determined by image scanning of randomly chosen photographs of the isolated fat cells. Skeletal muscle tissue will be obtained by percutaneous biopsy for histochemical determination of the fat content of muscle cells. A 75-g oral glucose tolerance test and a 25-g intravenous glucose tolerance test will be performed. Insulin action will be measured with a hyperinsulinemic-euglycemic glucose clamp (insulin infusion: 40mU/m(2) min) and insulin secretory responses to glucose will be measured during a 5-step hyperglycemic glucose clamp immediately thereafter. Pima subjects will be followed longitudinally after discharge from the unit and oral glucose tolerance tests will be performed every three months. Individuals who transition from normal to impaired glucose tolerance or impaired glucose tolerance to diabetic will be invited back to the Clinical Research Center for repeat testing.

By comparing insulin secretion-glucose dose-response curves, it may be possible to discern subtle defects in insulin secretion predisposing certain individuals to NIDDM. In addition, comparison of the responses in the offspring of diabetic pregnancies with those in the offspring of mothers who subsequently became diabetic may allow us to separate defects due to genetic causes from those due to the intrauterine environment. Finally, studying subjects as they progress from normal glucose tolerance to diabetes will test whether the defects in insulin secretion are progressive and contribute to the development of NIDDM.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy men and women (Pimas and non-Pimas)

At least 18 years of age

EXCLUSION CRITERIA:

Pregnancy and/or breastfeeding

Positive urine drug screening test

Inability to provide informed consent

Medical conditions or medications that, in the investigators' judgement, would affect glucose metabolism or insulin secretion. Examples include, but are not limited to: hyper- or hypothyroidism or other endocrine disorders, cardiovascular disease by history or examination, pancreatitis, hepatitis, cirrhosis or other gastrointestinal disease, renal insufficiency, active alcoholism or other substance abuse problems.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 1996-08-19; Study Completion 2011-08-16

CONTACTS AND LOCATIONS:
Locations (1):
- NIDDK, Phoenix, Phoenix, Arizona, United States

REFERENCES:
- [Background] Knowler WC, Pettitt DJ, Saad MF, Bennett PH. Diabetes mellitus in the Pima Indians: incidence, risk factors and pathogenesis. Diabetes Metab Rev. 1990 Feb;6(1):1-27. doi: 10.1002/dmr.5610060101. No abstract available. PMID 2192853
- [Background] Lillioja S, Mott DM, Zawadzki JK, Young AA, Abbott WG, Bogardus C. Glucose storage is a major determinant of in vivo "insulin resistance" in subjects with normal glucose tolerance. J Clin Endocrinol Metab. 1986 May;62(5):922-7. doi: 10.1210/jcem-62-5-922. PMID 3514652
- [Background] Lillioja S, Mott DM, Spraul M, Ferraro R, Foley JE, Ravussin E, Knowler WC, Bennett PH, Bogardus C. Insulin resistance and insulin secretory dysfunction as precursors of non-insulin-dependent diabetes mellitus. Prospective studies of Pima Indians. N Engl J Med. 1993 Dec 30;329(27):1988-92. doi: 10.1056/NEJM199312303292703. PMID 8247074
- [Derived] Koska J, Stefan N, Dubois S, Trinidad C, Considine RV, Funahashi T, Bunt JC, Ravussin E, Permana PA. mRNA concentrations of MIF in subcutaneous abdominal adipose cells are associated with adipocyte size and insulin action. Int J Obes (Lond). 2009 Aug;33(8):842-50. doi: 10.1038/ijo.2009.106. Epub 2009 Jun 9. PMID 19506561